CLINICAL TRIAL: NCT05034419
Title: Synaptic Plasticity in the Epicardial Ganglionated Plexi
Acronym: SNAP-GP
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of Oklahoma (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 11474
Record Dates: First submitted 2021-08-27; First posted 2021-09-05 (Actual); Last update posted 2024-03-06 (Actual); Status verified 2024-03

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Active stimulation (Experimental): Patients undergoing cardiac surgery will be randomized to active low level tragus stimulation for 30 min (pulse width of 200 μs, amplitude of 20 mA and a pulse frequency of 20 Hz). Stimulation will be provided using the Parasym device.
  Interventions: Device: Parasym
- Sham stimulation (Sham Comparator): Patients undergoing cardiac surgery will be randomized to sham stimulation for 30 min. The Parasym device will be placed on the patient's tragus, but no current will be delivered.
  Interventions: Device: Sham stimulation

INTERVENTIONS:
Device: Parasym — Stimulation will be done under anesthesia for 30 minutes. Stimulation parameters include a pulse width of 200 μs, amplitude of 20 mA and a pulse frequency of 20 Hz. The Parasym devise (Parasym Health, London, UK) will be used for stimulation. The device will be connected to a clip electrode that will be attached to the external ear. In the active group, the ear clip electrode will be attached to tragus in the active stimulation group. This device has been deemed non-significant risk by the FDA. In the control group, no stimulation will be done.
  Arms: Active stimulation
Device: Sham stimulation — Sham stimulation
  Arms: Sham stimulation

SUMMARY:
Atrial fibrillation (AF) is the most common arrhythmia and the prevalence increase with age. Autonomic nervous system play a critical role in the initiation and maintenance of AF. The intrinsic cardiac autonomic nervous system includes ganglionated plexus (GP) modulate the level of parasympathetic activity to the heart. Experimental and clinical studies suggest that GP activation plays a significant role in clinical AF in both the initiation of and the maintenance of AF.

Synaptic plasticity is defined as the ability of synapses to change their strength of transmission. Plasticity of synaptic connections in the brain is a major focus of neuroscience research, as it is the primary mechanism underpinning learning and memory. Beyond the brain however, plasticity in peripheral neurons is less well understood, particularly in the GP neurons innervating the heart. The ability of these neurons to alter parasympathetic activity suggests that plasticity may indeed occur at the synapses formed on and by GP neurons. Such changes may not only fine-tune autonomic innervation of the heart, but could also be a source of maladaptive plasticity during atrial fibrillation.

Low level tragus stimulation (LLTS) has been shown to decrease AF burden among patients with paroxysmal AF. However, the exact mechanism remains unclear. The objective of this study is to examine changes in synaptic density of GP neurons in patients with paroxysmal AF and persistent AF compared to those without AF undergoing cardiac surgery. In addition, we aim to examine the effect of LLTS on the synaptic plasticity of the GP neurons. A group of patients undergoing open heart surgery will be randomized to active LLTS for 30 min (pulse width of 200 μs, amplitude of 20 mA and a pulse frequency of 20 Hz) or no stimulation. Biopsy from GP tissue will be taken immediately after stimulation and histological staining for choline acetyl transferase (ChAT), tyrosine hydroxylase (TH) and synaptophysin will be performed to examine synaptic plasticity.

Understanding the effect of LLTS on GP SP will help to determine whether changes in synaptic plasticity can increase or decrease autonomic tone of the heart, and its role in generating the aberrant electrical impulses in the GP around the pulmonary veins that can trigger and drive AF.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female patients older than 21 year old
2. Patient is going to have open heart surgery.

Exclusion Criteria:

1. Patients undergoing emergent open heart surgery.

Ages: 21 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2021-03-24 (Actual); Primary Completion 2024-10 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
choline acetyltransferase | 30 minutes
  Biopsy from ganglionated plexus (GP) tissue will be taken and histological staining for choline acetyl transferase (ChAT) will be performed
tyrosine hydroxylase | 30 minutes
  Biopsy from ganglionated plexus (GP) tissue will be taken and histological staining for tyrosine hydroxylase will be performed
synaptophysin | 30 minutes
  Biopsy from ganglionated plexus (GP) tissue will be taken and histological staining for synaptophysin will be performed

CONTACTS AND LOCATIONS:
Locations (1):
- OU Medical Center, Oklahoma City, Oklahoma, United States

IPD SHARING:
Plan to Share IPD: Undecided